CLINICAL TRIAL: NCT00627341
Title: Addressing Fear of Food in Anorexia Nervosa
Brief Title: A Relapse Prevention Program for Reducing Relapse and Fear of Food in People With Anorexia Nervosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #5593; R01MH082736 (NIH); DATR A2-AID
Record Dates: First submitted 2008-02-28; First posted 2008-03-03 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Eating Disorders
Keywords: Exposure Therapy; Relapse Prevention; Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa | interventions — Secondary Prevention; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposure and Response Prevention (Experimental): Participants will receive Food Exposure Therapy and Ritual Prevention with Motivational Enhancement for Relapse Prevention in Anorexia Nervosa for 6 months.
  Interventions: Behavioral: Food Exposure Therapy and Ritual Prevention with Motivational Enhancement for Relapse Prevention in Anorexia Nervosa (AN-EX/RP)
- Cognitive Behavior Therapy (Active Comparator): Participants will receive cognitive behavioral therapy for anorexia nervosa for 6 months.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Food Exposure Therapy and Ritual Prevention with Motivational Enhancement for Relapse Prevention in Anorexia Nervosa (AN-EX/RP) — AN-EX/RP will consist of in-session exposures to feared eating situations without using avoidance behaviors as well as formal motivational interviewing techniques.
  Arms: Exposure and Response Prevention
Behavioral: Cognitive behavioral therapy (CBT) — CBT for anorexia nervosa sessions will focus on behaviorally normalizing eating patterns throughout the day and on cognitively addressing dysfunctional thinking that promotes disordered eating.
  Arms: Cognitive Behavior Therapy

SUMMARY:
This study will compare the effectiveness of two types of psychotherapy, a relapse prevention program and cognitive behavioral therapy, in reducing relapse and fear of eating situations in people with anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious and often chronic eating disorder characterized by restrictive eating habits and failure to maintain a healthy minimal body weight. Symptoms of AN may include distorted body image, fear of weight gain, obsessive exercise, and binge and purge eating behaviors. In severe cases of AN, a person may practice extreme dieting to levels of near starvation. These unhealthy behaviors may cause further medical complications, including organ damage, irregular heart rhythm, premature osteoporosis, and heart failure. AN has one of the highest mortality rates of all psychiatric disorders, claiming the lives of up to 6% of those affected. When treated with a form of psychotherapy and nutritional guidance, people can restore weight to healthy levels and recover from AN, but the chance of relapse remains high. A program aimed specifically at reducing relapse, Exposure Therapy and Ritual Prevention with Motivational Enhancement for Relapse Prevention in Anorexia Nervosa (AN-EX/RP), may be more effective than common psychotherapy treatments, such as cognitive behavioral therapy (CBT), in enhancing long-term recovery from AN. This study will compare the effectiveness of AN-EX/RP with CBT in reducing relapse and fear of eating situations in people with AN.

Participants in this study will include patients who have achieved normal weight while inpatients at the New York State Psychiatric Unit. Eligible participants will undergo initial assessments that will include questionnaires, interviews, and two laboratory-based meals. Participants will then be assigned randomly to receive 6 months of outpatient psychotherapy treatment with either AN-EX/RP or CBT. Participants assigned to receive AN-EX/RP will attend 90-minute sessions twice weekly for the first few months, then weekly thereafter. Sessions will focus on fear of eating situations and will help participants to confront, rather than avoid, these fears in order to learn through practice that the fears are unrealistic. Participants assigned to receive CBT will attend treatment sessions twice weekly for the first month and then weekly thereafter. CBT sessions will focus on thoughts, feelings, and behaviors that perpetuate the eating disorder, with the aim to develop healthier patterns. After completing the 6 months of treatment, all participants will repeat the initial assessments.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV-TR criteria for anorexia nervosa (restricting or binge-purge subtype), with or without amenorrhea after inpatient admission
* Has achieved 90% of ideal body weight or BMI greater than or equal to 19.5 kg/m2 for at least 1 week after inpatient admission
* Medically stable

Exclusion Criteria:

* Chronic psychotic or bipolar I disorder requiring ongoing treatment with antipsychotic or mood stabilizer
* Diagnosis of obsessive compulsive disorder in which the symptoms are clearly unrelated to eating disorders
* Current substance abuse
* Current use of psychotropic medication
* Acute suicidality (suicidality or self-injury in the 3 months before study entry)
* Serious medical illness

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Diet Energy Density and Variety score | Measured before treatment and at Months 1, 2, 3, 4, 5, and 6

SECONDARY OUTCOMES:
Yale-Brown-Cornell Obsessive-Compulsive Scale for Eating Disorders (YBC-EDS) score | Measured before treatment and at Months 3 and 6
Body mass index (BMI) | Measured weekly for 6 months
Amount consumed at test meals | Measured two times before treatment and two times after Month 6
Reported levels of anxiety at test meals | Measured two times before treatment and two times after Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Joanna E. Steinglass, MD, Principal Investigator — Research Foundation for Mental Hygiene, Inc.
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Steinglass JE, Albano AM, Simpson HB, Wang Y, Zou J, Attia E, Walsh BT. Confronting fear using exposure and response prevention for anorexia nervosa: A randomized controlled pilot study. Int J Eat Disord. 2014 Mar;47(2):174-80. doi: 10.1002/eat.22214. Epub 2013 Nov 8. PMID 24488838
- [Derived] Steinglass JE, Sysko R, Mayer L, Berner LA, Schebendach J, Wang Y, Chen H, Albano AM, Simpson HB, Walsh BT. Pre-meal anxiety and food intake in anorexia nervosa. Appetite. 2010 Oct;55(2):214-8. doi: 10.1016/j.appet.2010.05.090. Epub 2010 Jun 4. PMID 20570701